CLINICAL TRIAL: NCT03840395
Title: The PhINEST Study - Pharyngeal ICU Novel Electrical Stimulation Therapy: a Prospective, Multi-site, Randomised, Sham-controlled, Single-blind (outcome Assessor-blinded) Study.
Brief Title: The PhINEST Study - Pharyngeal ICU Novel Electrical Stimulation Therapy
Acronym: PhINEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Phagenesis Ltd. (Industry)
Collaborators: NAMSA (Other); Cytel Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHE-06
Record Dates: First submitted 2019-01-30; First posted 2019-02-15 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Dysphagia
Keywords: Dysphagia; Extubation; Intensive Care Unit; Pharyngeal Electrical Stimulation; Oropharyngeal Dysphagia; Mechanical Ventilation; Critically ill patients; Post-Extubation Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active PES (Active Comparator): Patients randomized to receive active Pharyngeal Electrical Stimulation (PES) via a Phagenyx Catheter.
  Interventions: Device: Pharyngeal Electrical Stimulation (PES)
- Sham PES (Sham Comparator): Patients randomized to sham will not receive any Pharyngeal Electrical Stimulation (PES) but will still have the Phagenyx Catheter inserted.
  Interventions: Device: Pharyngeal Electrical Stimulation (PES)

INTERVENTIONS:
Device: Pharyngeal Electrical Stimulation (PES) — The Phagenyx® system is a two-part neurostimulation system. It is composed of a durable component called the Base Station and the single-use sterile disposable Catheter. The Base Station acts as the user interface and provides the means to generate, optimize and monitor the delivery of electrical stimulation to the oropharynx. The Phagenyx® devices are CE labelled (2012) and will be used in accordance with their intended use label.
  Other Names: Phagenyx

SUMMARY:
This is a prospective, multi-site, randomised, sham-controlled, single-blind (outcome assessor-blinded) study designed to assess the effects of Pharyngeal Electrical Stimulation (PES) (using Phagenyx®) for the treatment of oropharyngeal dysphagia after invasive mechanical ventilation (of any duration) by means of naso or oro-tracheal tube in critically ill intensive care unit (ICU) patients.

DETAILED DESCRIPTION:
The PhINEST study is designed to assess the effects of Pharyngeal Electrical Stimulation (PES) (using Phagenyx®) for treatment of oropharyngeal dysphagia after invasive mechanical ventilation (of any duration) by means of naso or oro-tracheal tube in critically ill intensive care unit (ICU) patients.

The main clinical outcomes assessing unsafe swallows and dysphagia severity will be measured using the gold standard, i.e. Fiberoptic Endoscopic Evaluation of Swallowing (FEES) and bedside swallowing assessments on day 2* after completion of final PES treatment.

Randomisation will be on a 1:1 basis at each site stratified for neurological vs. non-neurological reason for admission (Acute Physiology and Chronic Health Evaluation (APACHE) IV diagnostic group). Patients will receive either PES/sham treatment in addition to standard supportive ICU care and standard of care treatments for dysphagia. Administration of all protocol-specific assessments will be conducted by personnel blinded to treatment assignment.

The study will follow an adaptive population enrichment and sample size re-estimation (SSR) design with one interim look. The study will start with a planned sample size of 200 patients and a maximum (evaluable) sample size of 360. Interim analysis after completion of approximately 140 (evaluable) patients will determine:

I. futility stopping; OR II. sample size increase for the overall sampled population; OR III. Enrichment based on the composite primary endpoint by pre-defined subgroups (neurological vs. non-neurological reason for admission according to APACHE IV diagnostic groups). Thus enrollment of patients in the non-performing sub-group will be stopped at the interim while a sample-size re-estimation based on conditional power will be carried out for the other sub-group.

All interim decisions will be based on conditional power which for the Finkelstein-Schoenfeld (FS)-statistic will need to be computed via Monte-Carlo simulations.

Up to thirty (30) investigational sites across Europe are planned to participate in this study which is expected to last 48 months from first patient first visit to last patient last visit. Patients will be assessed at the following intervals: screening, baseline, on day 2* after completion of final study treatment, 7 ± 1 days after final study treatment and 14 ± 1 days after final study treatment (or hospital discharge if earlier). 30-day and 90-day mortality data will also be collected from the patients medical notes/electronic heath records/telephone call (no additional visit required).

*The day two (FU1) visit is to be conducted on the second day (~24hrs) following final PES treatment but may, under certain circumstances, be conducted upon/by the fourth day (~60 hrs) following final study treatment in instances where the final study treatment is delivered on late Friday and where FEES assessment is only possible early on Monday as no weekend FEES service is available at the investigation site.

ELIGIBILITY:
Pre-screening Inclusion Criteria:

All of the following criteria must be met for inclusion:

* Age ≥ 18 ≤ 85,
* Emergency ICU admission (unplanned admission),
* Recent extubation following invasive mechanical ventilation (of any length of time) by means of endotracheal tube,
* Presence of post-extubation dysphagia as determined by the participating Sites' Standard Of Care (SOC).

Screening / Enrolment Criteria:

To be eligible for enrolment in this study, an individual must meet all of the following additional criteria:

* Presence of written informed consent according to respective national guidelines,
* Dysphagia severity status classified according to PAS on FEES assessment as 'aspiration' (PAS score ≥ 6),
* Richmond Agitation and Sedation Scale (RASS) score within the range of -1 to +2 (i.e. if score equals -2, -3, -4 or +3, +4, patient is excluded).

Randomisation Inclusion Criteria (post-consent)

The following additional criteria must be met for randomisation:

• Successful placement and subjective tolerance of the Phagenyx® Catheter within 2 days of extubation.(post consent)

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from enrolment in this study:

* Nasal anatomical deformity, nasal airway obstruction; patient who have had recent oral, nasal or oesophageal surgery or patient presenting with facial and/or cranial fractures or any other circumstance (e.g. history of oesophageal perforation, stricture, pouch, resection or rupture) where the placement of a standard nasogastric feeding tube (NGT) would be deemed unsafe,
* Cardiac or respiratory condition that might render the insertion (placement) of a catheter into the throat unsafe,
* Permanently implanted electrical devices,
* Are pregnant (pregnancy test) or known lactating women,
* Have non-neurogenic dysphagia (e.g. Cancer-related),
* Any prior tracheostomy,
* Patients who at the time of extubation have any treatment limitation (i.e., palliative care, life expectancy less than 48 hours, or are moribund), that prevents or would prevent compliance with study-specific instructions or procedures (as judged by the investigator),
* Severe cognitive impairment or other reasons that prevents compliance with study-specific instructions or procedures (as judged by the investigator),
* Previous history of dysphagia of any origin,
* Pre-existing tube feeding of any form (e.g. percutaneous gastric/enteral feeding tube related to previous injuries indicating previous dysphagia. NGTs are not an exclusion criterion),
* Participation in another interventional study (medicinal or device) that could influence the outcomes of PES,
* Treatment of dysphagia with other forms of electrical stimulation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Phagenyx® treatment in reducing severity of unsafe swallows - Penetration-Aspiration Scale (PAS) Scores | Day 2 (~24 to ~60 hours) after the final Phagenyx® treatment
  Analysis of a two endpoints composite (FS-statistic) on a hierarchy of clinical priorities:
  Endpoint 1 - Swallowing safety based on worst PAS score in up to 4 thin (water) boli for each patient during FEES assessment converted to a trichotomised ordinal response of safe (PAS 1-3), penetration (PAS 4-5), or aspiration (PAS 6-8).
  The PAS provides a scoring system for airway closure and clearance during FEES. The PAS is a validated 8-point scale quantifying penetration and aspiration events primarily by the depth to which material passes into the airway and whether or not it is ejected.
Effectiveness of Phagenyx® treatment in reducing the severity of unsafe swallows - Dysphagia Outcome and Severity Score (DOSS) score | 7±1 days after the final Phagenyx® treatment
  Analysis of a two endpoints composite (FS-statistic) on a hierarchy of clinical priorities:
  Endpoint 2 - DOSS scale score determined by bedside assessment.
  The DOSS is a simple, easy-to-use, 7-point scale developed to systematically rate the functional severity of dysphagia based on objective assessment and make recommendations for diet level, independence level, and type of nutrition.
  1. Severe dysphagia
  2. Moderately severe dysphagia
  3. Moderate dysphagia
  4. Mild-moderate dysphagia
  5. Mild dysphagia
  6. Functional limitation and modified independence
  7. Normal in all situations

SECONDARY OUTCOMES:
Effectiveness of Phagenyx® treatment in improving DOSS score. | Up to 14 ± 1 days after the final Phagenyx® treatment (or hospital discharge if earlier).
  Changes in nutritional management and severity of dysphagia as measured by the DOSS score.
Effectiveness of Phagenyx® treatment on time from to feeding tube removal. | Up to 14 ± 1 days after the final Phagenyx® treatment (or hospital discharge if earlier).
  Changes in nutritional management and severity of dysphagia as measured by time from randomisation to removal of feeding tube.
Effectiveness of Phagenyx® treatment on time to oral intake. | Up to 14 ± 1 days after the final Phagenyx® treatment (or hospital discharge if earlier).
  Changes in nutritional management and severity of dysphagia as measured by time to oral intake (if applicable).
Effectiveness of Phagenyx® treatment on total days of enteral feeding. | Up to 14 ± 1 days after the final Phagenyx® treatment (or hospital discharge if earlier).
  Changes in nutritional management and severity of dysphagia as measured by total days of enteral feeding.
Effectiveness of Phagenyx® treatment in improving Functional Oral Intake Scale (FOIS) score. | Up to 14 ± 1 days after the final Phagenyx® treatment (or hospital discharge if earlier).
  Changes in nutritional management and severity of dysphagia as measured by the FOIS score.
  The FOIS provides a scoring system to document the functional level of oral intake of food and liquid in patients with dysphagia. It is a validated 7-point ordinal scale easily completed from information contained in medical charts, dietary journals, and/or patient reports.
  1. Nothing by mouth
  2. Tube dependent with minimal attempts of food or liquid
  3. Tube dependent with consistent intake of liquid or food
  4. Total oral diet of a single consistency
  5. Total oral diet with multiple consistencies but requiring special preparation or compensations
  6. Total oral diet with multiple consistencies without special preparation, but with specific food limitations
  7. Total oral diet with no restriction
Effectiveness of Phagenyx® treatment in improving Dysphagia Severity Rating Scale (DSRS) score. | Up to 14 ± 1 days after the final Phagenyx® treatment (or hospital discharge if earlier).
  Changes in nutritional management and severity of dysphagia as measured by the DSRS score.
  The DSRS is a simple to use, validated 13-point scale composed of a 3-component score that includes feeding independence, but nutrition level and diet modification is split into the components of liquid feeding and overall diet consistency. The DSRS is the sum of the scores of each of the 3 individual components (range 0-4 for each component) rather than a combination of the three components into an ordinal scale.
  Best score = 0 (no dysphagia) Worst score = 12 (NPO)
Effectiveness of Phagenyx® treatment on time from extubation to ICU discharge | Up to 14 ± 1 days after the final Phagenyx® treatment (or hospital discharge if earlier).
  General health outcome measured by time from extubation to ICU discharge (days).
Effectiveness of Phagenyx® treatment on length of stay in ICU | Up to 14 ± 1 days after the final Phagenyx® treatment (or hospital discharge if earlier).
  General health outcome measured by length of stay in ICU (days).
Effectiveness of Phagenyx® treatment on length of stay in hospital. | Up to 14 ± 1 days after the final Phagenyx® treatment (or hospital discharge if earlier).
  General health outcome measured by length of stay in hospital (days).
Effectiveness of Phagenyx® treatment on number of patients with re-intubation during hospital stay | Up to 14 ± 1 days after the final Phagenyx® treatment (or hospital discharge if earlier).
  General health outcome measured by number of patients with re-intubation during hospital stay.
Effectiveness of Phagenyx® treatment on mortality | Up to 90 days after completion of the final Phagenyx® treatment.
  General health outcome measured by 30-day and 90-day mortality.

OTHER OUTCOMES:
Effectiveness of Phagenyx® treatment in reducing (dysphagia) secretion severity. | Day 2 (~24 to ~60 hours) after the final Phagenyx® treatment
  Exploratory analysis of changes in secretion severity (severity of dysphagia) between FEES assessments measured by an Independent FEES Review Committee (IFRC) using the Murray Secretion Severity Rating Scale (SSS).
  The SSS is a simple, easy-to-use, 4-point scale that can systematically rate the graduation of accumulated secretions within the pharyngolarynx and trachea during FEES.
  0. Normal
  1. Mild
  2. Moderate
  3. Severe
Effectiveness of Phagenyx® treatment in improving swallowing safety and efficiency - PAS scores | Day 2 (~24 to ~60 hours) after the final Phagenyx® treatment
  Exploratory analysis of changes in swallowing safety and efficiency (severity of dysphagia) between FEES assessments measured by an IFRC based on worst PAS score for each bolus consistency (semi-solid and solid) for each patient during FEES assessment converted to a dichotomised ordinal response of non-aspirator (PAS 1-5) or aspirator (PAS 6-8).
Effectiveness of Phagenyx® treatment in reducing bolus residue | Day 2 (~24 to ~60 hours) after the final Phagenyx® treatment
  Exploratory analysis of changes in bolus residue (severity of dysphagia) between FEES assessments measured by an IFRC using the Yale Pharyngeal Residue Severity Rating Scale (YRS).
  The YRS is a reliable, validated, anatomically defined, and image-based five-point ordinal rating scale to determine severity of post-swallow pharyngeal residue location (vallecula and pyriform sinus) and amount (i. none, ii. trace, iii. mild, iv. moderate, and v. severe) during FEES.
Effectiveness of Phagenyx® treatment in reducing global dysphagia severity | Day 2 (~24 to ~60 hours) after the final Phagenyx® treatment
  Exploratory analysis of changes in severity of dysphagia between FEES assessments measured by an IFRC using the Global Dysphagia Severity Rating Scale (GDS).
  The GDS is a simple, easy-to-use, 4-point scale developed to systematically rate the severity of dysphagia during FEES.
  0. No relevant dysphagia
  1. Mild dysphagia: Premature spillage and/or residues, but no penetration/aspiration events.
  2. Moderate dysphagia: Penetration/aspiration events with one consistency.
  3. Severe dysphagia: Penetration/aspiration events with two or more consistencies.
Effectiveness of Phagenyx® treatment on time from extubation to hospital discharge | Up to 14 ± 1 days after the final Phagenyx® treatment (or hospital discharge if earlier).
  Exploratory analysis of general health outcome measured by time from extubation to hospital discharge (days).
Effectiveness of Phagenyx® treatment on days on antimicrobials post-extubation (while in ICU) | Up to 14 ± 1 days after the final Phagenyx® treatment (or hospital discharge if earlier).
  Exploratory analysis of general health outcome measured by days on antimicrobials post-extubation (while in ICU).
Effectiveness of Phagenyx® treatment on hospital discharge destination | Up to 90 days after the final Phagenyx® treatment
  Exploratory analysis of general health outcome measured by hospital discharge destination (home, home+care, nursing home, other hospital, rehabilitation centre).
Effectiveness of Phagenyx® treatment on ICU readmission rate during hospital stay | Up to 14 ± 1 days after the final Phagenyx® treatment (or hospital discharge if earlier).
  Exploratory analysis of general health outcome measured by ICU readmission rate during hospital stay.
Effectiveness of Phagenyx® treatment on tracheostomies per subgroup | Up to 14 ± 1 days after the final Phagenyx® treatment (or hospital discharge if earlier).
  Exploratory analysis of general health outcome measured by number of and reason for tracheostomies per subgroup after PES-treatment during hospital stay.
Effectiveness of Phagenyx® treatment on chest X-rays for suspected pneumonia. | Up to 14 ± 1 days after the final Phagenyx® treatment (or hospital discharge if earlier).
  Exploratory analysis of general health outcome measured by total number of chest X-rays during hospital stay after ICU discharge for suspected pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Schefold, MD, Principal Investigator — University Clinic for Intensive Medicine, Inselspital, University of Bern; Micheal Joannidis, MD, Principal Investigator — Medizinische Universität Innsbruck - Universitätsklinik für Innere Medizin I; Christopher Rugg, MD, Principal Investigator — Medizinische Universität Innsbruck - Universitätsklinik für Anästhesie und Intensivmedizin; Alois Schiefecker, MD, Principal Investigator — Medizinische Universität Innsbruck - Universitätsklinik für Neurologie; Stefan Kluge, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf - Klinik für Intensivmedizin
Locations (7):
- Austria (3):
  - Medizinische Universität Innsbruck - Medizinische Universität Innsbruck, Innsbruck
  - Medizinische Universität Innsbruck - Universitätsklinik für Anästhesie und Intensivmedizin, Innsbruck
  - Medizinische Universität Innsbruck - Universitätsklinik für Innere Medizin I, Innsbruck
- Finland (2):
  - Helsinki University Hospital Perioperative, Intensive Care and Pain Medicine, Helsinki
  - Oulu University Hospital, Oulu
- Universitätsklinikum Hamburg-Eppendorf - Klinik für Intensivmedizin, Hamburg, Germany
- University Clinic for Intensive Medicine, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schefold JC, Backlund M, Ala-Kokko T, Zuercher P, Mukherjee R, Mistry S, Mayer SA, Dziewas R, Bakker J, Jakob SM. The PhINEST study - Pharyngeal ICU Novel Electrical Stimulation Therapy: Study protocol of a prospective, multi-site, randomized, sham-controlled, single-blind (outcome assessor-blinded) study. Medicine (Baltimore). 2020 Mar;99(11):e19503. doi: 10.1097/MD.0000000000019503. PMID 32176093
- [Derived] Likar R, Aroyo I, Bangert K, Degen B, Dziewas R, Galvan O, Grundschober MT, Kostenberger M, Muhle P, Schefold JC, Zuercher P. Management of swallowing disorders in ICU patients - A multinational expert opinion. J Crit Care. 2024 Feb;79:154447. doi: 10.1016/j.jcrc.2023.154447. Epub 2023 Nov 2. PMID 37924574
- See also: PhINEST Study - Protocol Manuscript — https://pubmed.ncbi.nlm.nih.gov/32176093/